CLINICAL TRIAL: NCT02307695
Title: The Effect of Saxagliptin on Glucose Fluctuation and Immune Regulation in Patients With Type 1 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yang Tao, Department of Endocrinology & Metabolism, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-SR-123
Record Dates: First submitted 2014-11-12; First posted 2014-12-04 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Type 1 Diabetes
Keywords: Saxagliptin; Type 1 Diabetes; Glycemic variability; C-Peptide
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — saxagliptin; Dipeptidyl-Peptidase IV Inhibitors; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- insulin+Saxagliptin (Experimental): Patients who have diagnosed type 1 diabetes are assigned to receive Saxagliptin tablets 5 mg and insulin for 24-week.
  Interventions: Drug: Saxagliptin; Drug: Insulin
- insulin (Active Comparator): Patients who have diagnosed type 1 diabetes only use insulin.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Saxagliptin — saxagliptin 5 mg p.o. qd, 24 week
  Other Names: Onglyza; DPP-IV inhibitor
  Arms: insulin+Saxagliptin
Drug: Insulin — Patients will be treated according to routine clinical practice at the discretion of the treating physician.

SUMMARY:
To investigate whether saxagliptin could reduce the fluctuation of glycemia and improve the glycemic control in those type 1 diabetes through mechanisms of suppressing glucagon secretion, improving beta cell function, and re-regulating of the T cell immune system.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) is characterized by immune mediated beta-cell destruction. Due to the imbalance between glucagon and insulin, long-term T1DM patients experience frequent hypoglycaemia and high glucose variability despite of multiple daily injections of insulin.

Dipeptidyl peptidase 4 (DPP-4) inhibitors are a new class of anti-diabetic agents and are widely used in clinical practice to improve glycemic control and protect β-cell function in patients with type 2 diabetes mellitus(T2DM). Saxagliptin, a DPP-4 inhibitor, improves glycemic control in patients with T2DM by increasing endogenous active, intact glucagon-like peptide 1 and glucose-dependent insulinotropic polypeptide in response to food, which augments insulin secretion and decreases glucagon release. This mechanism can lead to the reduction of glucose variation. In some pilot studies, incretin-based therapy in patients with T1DM can improve glucose control and reduce hypoglycemia, the mechanism probably is that it regulates glucagon level. In type 1 diabetic mouse models, DPP-4 inhibitors preserves beta-cell mass and stimulating beta-cell replication.

Interestingly, DPP-4 is also known as cluster of differentiation antigen 26(CD26).It is expressed on the membrane of many types of lymphocyte, e.g. T, B and natural killer(NK)cells, and is involved in their cellular functions. CD26 plays a key role in many aspects in lymphocyte function beyond its DPP-4 enzymatic activity.These observations make it a promising therapeutic target.

Recently, the attention of saxagliptin has been mainly focused on type 2 diabetes, data in type 1 diabetes is rare. We are going to carry out this phase 4 study to testify our hypothesis that saxagliptin could reduce the fluctuation of glycemia and improve the glycemic control in those type 1 diabetes through mechanisms of suppressing glucagon secretion, improving beta cell function, and re-regulating of the T cell immune system.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures;
2. Diagnosed with type 1 diabetes;
3. Men or women who are 12 to 65 years of age at time of consenting upon Visit 1.;
4. Positivity for at least one of the four islet autoantibodies(IA-2A、IAA、GADA、ZnT8A);
5. 6.5% ≤ HbA1c ≤10.0%.

Exclusion Criteria:

1. type 2 diabetes；
2. Evidence of chronic or acute complications of diabetes which is unstable and requires hospitalization；
3. Evidence of disease stress；
4. History of administration of any antihyperglycemic therapy (other than insulin) during the 12 weeks prior to Visit 1；
5. Have a history of, or currently have, acute or chronic pancreatitis；
6. Immunocompromised individuals such as patients that have undergone organ transplantation or patients diagnosed with HIV or patients with agranulocytosis；
7. Evidence of chronic or acute infection；
8. Active liver disease and/or significant abnormal liver function defined as Aspartate transaminase(AST) ≥3x Upper Limit of Normal(ULN) and/or Alanine aminotransferase (ALT) ≥3x Upper Limit of Normal(ULN)；
9. History of unstable or rapidly progressing renal disease, creatinine clearance(CrCl) ≤50ml/min;
10. Congestive heart failure defined as New York Heart Association (NYHA) class III or IV and/or left ventricular ejection fraction of ≤ 40%；
11. Rheumatoid arthritis or other autoimmune disease(except AITD);
12. Hypersensitivity to saxagliptin；
13. History of drug allergy or allergic disease
14. History of alcohol abuse, illegal drug abuse, mental disease or other disease which is not eligible for the study
15. Pregnant or breastfeeding patients；
16. Patients with any diseases which in the judgement of the investigator would compromise the patient's safety or successful participation in the clinical study
17. Any condition where, in the opinion of the investigator, participation in this study may pose a significant risk to the patient or could render the patient unable to successfully complete the study
18. Any disease or condition which the investigator feels would interfere with the trial;
19. Treatment with other immunosuppressive agent such as systemic glucocorticoids other than replacement therapy. Inhaled, local injected and topical use of glucocorticoids is allowed during the last 90 days prior to Visit 1;
20. Participation in a clinical study during the last 90 days prior to Visit 1;
21. Patients who are participating in other clinical study;
22. Treatment with strong cytochrome P450 3A4/5 (CYP3A4/5) inhibitors or other contraindications to therapy as outlined in the saxagliptin package insert;
23. History of haemoglobinopathies (sickle cell anaemia or thalassemias, sideroblastic anaemia).

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change of Mean amplitude of glycemic excursions (MAGE) from baseline in patients with type 1 diabetes treated with saxagliptin plus insulin or insulin alone by continuous glucose monitoring system (CGMS) | 24 week

SECONDARY OUTCOMES:
Change of C-peptide area under the curve (AUC C-peptide) or fasting C-peptide from baseline in patients with type 1 diabetes treated with saxagliptin plus insulin or insulin alone by 3-hour mixed meal tolerance test(MMTT) | 24 week
Change of Haemoglobin A1c (HbA1c) from baseline in patients with type 1 diabetes treated with saxagliptin plus insulin or insulin alone | 24 week
Change of insulin dosage (U/kg/d) from baseline in patients with type 1 diabetes treated with saxagliptin plus insulin or insulin alone | 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yang, MD/PhD, Principal Investigator — First Affiliated Hospital, Nanjing Medical University, China
Locations (1):
- First Affiliated Hospital, Nanjing Medical University, Nanjing, Jiangsu, China